CLINICAL TRIAL: NCT02429271
Title: A Multicenter Trial to Assess the MIcrovascular Integrity and Left Ventricular Function Recovery After Clopidogrel or TicagrelOr Administration, in Patients With STEMI Treated With Thrombolysis - The 'MIRTOS' Study
Acronym: MIRTOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hellenic Cardiovascular Research Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D5130C00137
Record Dates: First submitted 2015-04-17; First posted 2015-04-29 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Myocardial Infarction; ST Segment Elevation Myocardial Infarction (STEMI)
Keywords: undergoing thrombolysis
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — Ticagrelor; Clopidogrel; Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Active Comparator): 1st day 270 mg & from then onwards 180 mg per day
  Interventions: Drug: Ticagrelor; Procedure: Percutaneous Coronary Intervention (PCI); Procedure: Coronary Angiography
- Clopidogrel (Active Comparator): 1st day 300 mg & from then onwards 75 mg per day
  Interventions: Drug: Clopidogrel; Procedure: Percutaneous Coronary Intervention (PCI); Procedure: Coronary Angiography

INTERVENTIONS:
Drug: Ticagrelor
  Other Names: Brilique
  Arms: Ticagrelor
Drug: Clopidogrel
  Other Names: Plavix
  Arms: Clopidogrel
Procedure: Percutaneous Coronary Intervention (PCI)
Procedure: Coronary Angiography

SUMMARY:
This is a prospective randomized study, which investigates the coronary microvascular function as assessed by coronary angiography after administration of ticagrelor compared with clopidogrel in patients with myocardial infarction and ST segment elevation after thrombolysis.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Male and female subjects, 18-75 years of age (both inclusive).
3. STEMI eligible for thrombolysis
4. Inability to perform primary PCI, because of transport time in centers carrying out primary PCI lasting more than two hours
5. Ability of transportation in 3-24 hours after thrombolysis in order to perform coronary angiography and PCI. This period may be extended for reasons of extreme importance up to 72 hours at the latest.

Exclusion Criteria:

1. Inability to give informed consent.
2. Pre-treatment with any inhibitor of the purinergic receptor P2Y, G-protein coupled, 12 (P2Y12) within the 7-day period prior to randomization.
3. Cardiogenic shock - according to Killip classification - class 4.
4. Suspicion or evidence of mechanical complication, including mitral valve dysfunction, ventricular septal rupture, and rupture of the left ventricle.
5. Current use of warfarin or other anticoagulant drug.
6. Known multivessel coronary artery disease not suitable for revascularization.
7. Any contraindication to thrombolytic therapy -Central nervous system damage or neoplasms or atrioventricular malformation -Recent major trauma/surgery/head injury (within the preceding 3 weeks) -Gastrointestinal bleeding within the past month -Known bleeding disorder (excluding menses) -Aortic dissection -Non-compressible punctures in the past 24 hours (e.g. liver biopsy, lumbar puncture).
8. Other bleeding diathesis, or considered by Investigator to be at high risk for bleeding.
9. Any kind of stroke in the past year or haemorrhagic stroke ever.
10. Severe uncontrolled hypertension (>180/110 mmHg) prior to randomisation.
11. Prolonged or traumatic cardiopulmonary resuscitation (> 10 minutes) in the last 2 weeks.
12. Known thrombocytopenia defined as platelet count of <100,000/mm3.
13. Known anemia (hemoglobin [Hb] <10 gr/dL).
14. Subjects receiving daily treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase-2 (COX-2) inhibitors that cannot be discontinued for the duration of the study.
15. Chronic dialysis or known chronic renal failure (glomerular filtration rate (GFR)<30 ml/min/1.73m2).
16. Known moderate or severe hepatic impairment.
17. Severe uncontrolled chronic obstructive pulmonary disease.
18. Concomitant use of potent Cytochrome P450 3A4 (CYP3A4) inhibitors (atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin and voriconazole, grapefruit juice over 1 litre daily), CYP3A substrates with narrow therapeutic indices (cyclosporine, quinidine), or inducers (carbamazepine, dexamethasone, phenobarbital, phenytoin, rifampin, and rifapentine).
19. Concomitant use of drugs that are metabolized through cytochrome P450, family 2, subfamily C, polypeptide 19 (CYP2C19) (omeprazole and esomeprazole, fluvoxamine, fluoxetine, moclobemide, voriconazole, fluconazole, ticlopidine, ciprofloxacin, cimetidine, carbamazepine, oxcarbazepine and chloramphenicol).
20. Increased risk of bradycardic events (e.g. known sick sinus syndrome or third degree atrioventricular (AV) block or previous documented syncope suspected to be due to bradycardia unless treated with a pacemaker).
21. Any known contraindication to clopidogrel, Acetylsalicylic Acid (ASA), or ticagrelor.
22. Current pregnancy, active lactation or parturition (childbirth) within the previous 30 days; women of childbearing potential must have a negative urine pregnancy test, or use a medically accepted method of birth control.
23. Treatment with other investigational agents (including placebo) or devices within 30 days prior to randomization or planned use of investigational agents or devices prior to the completion of study participation.
24. Any non-cardiac condition with life expectancy less than 1 year.
25. Inability to adhere to the follow-up requirements or any other reason or condition that the investigator feels would place the patient at increased risk if the investigational therapy is initiated.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2015-08; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
The difference in Post PCI Corrected TIMI Frame Count (CTFC) between the ticagrelor and clopidogrel treatment arms. | 15 months after the initiation of the study.

SECONDARY OUTCOMES:
The rates of TIMI Myocardial Perfusion Grade (TMPG) and the difference in the incidence of normal TMPG (3) following PCI between the ticagrelor and clopidogrel treatment arms. | 15 months after the initiation of the study.
The rates of Pre and Post PCI TIMI Flow Grade (TFG) and the difference in the incidence normal epicardial flow (TFG 3) following PCI between the ticagrelor and clopidogrel treatment arms. | 15 months after the initiation of the study.
The rates of full, partial and failed perfusion as assessed by the Angiographic Perfusion Score (APS) and the between treatment difference. | 15 months after the initiation of the study.
The rates of Thrombolysis In Myocardial Infarction (TIMI) thrombus grades Pre and Post PCI and the difference in the incidence of thrombus grade '0' following PCI between the ticagrelor and clopidogrel treatment arms. | 15 months after the initiation of the study.
The mean Global Longitudinal Strain (GLS) and Regional Longitudinal Strain (RLS) within 48 hours and at 30 and 90 days following PCI in the ticagrelor and clopidogrel treatment arms, and the between treatment difference. | 15 months after the initiation of the study.
The mean Left Ventricular Ejection Fraction (LVEF) within 48 hours and at 30 and 90 days following PCI in the ticagrelor and clopidogrel treatment arms, and the between treatment difference. | 15 months after the initiation of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Heraklion Venizeleio-Pananeio, Heraklion, Crete, Greece

REFERENCES:
- [Derived] Hamilos M, Kanakakis J, Anastasiou I, Karvounis C, Vasilikos V, Goudevenos J, Michalis L, Koutouzis M, Tsiafoutis I, Raisakis K, Stakos D, Hahalis G, Vardas P; Collaborators. Ticagrelor versus clopidogrel in patients with STEMI treated with thrombolysis: the MIRTOS trial. EuroIntervention. 2021 Feb 19;16(14):1163-1169. doi: 10.4244/EIJ-D-20-00268. PMID 32715996